CLINICAL TRIAL: NCT06590376
Title: The Effect of Midwifery Care Based on Swanson Care Theory Given to Couples Experiencing Pregnancy Loss on the Level of Grief and General Well-Being
Brief Title: The Effect of Midwifery Care Given to Couples Experiencing Pregnancy Loss on Grief and General Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Uskudar University (Other)
Responsible Party: Principal Investigator, Ayça Demir Yıldırım, PhD, Assistant Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ÜskudarU Betül Altay; BETÜL ALTAY (Other: USKUDARU)
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Pregnancy Loss; Grief; Loss Pregnancy; Care Pattern, Maternal; Bereavement
Keywords: Midwifery; pregnancy loss; perinatal bereavement; bereavement care guide; midwifery care and counselling

STUDY DESIGN:
Intervention Model Description: The research was designed as a randomized controlled, 2-group (intervention and control) pre-test post-test comparative experimental research.
Who Masked: Participant
Masking Description: The numbers from 1 to 96 were randomly allocated into two groups on the random.org website and randomly selected numbers were assigned to the intervention and control groups. This process ensured that the participants were equally and randomly distributed to the intervention and control groups. The group to which the case would be assigned was determined according to the order of hospitalisation and recorded in the Excel list.
  Since the care intervention and data collection in the study were carried out by the researcher, one-way blinding was performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Intervention group (Group receiving midwifery care based on Swanson Care Theory) (Experimental): After randomization of the women who were allocated to the clinic, they were informed about the research and their consent was obtained; then, the Women's Introductory Information Form, General Well-Being Scale, Perinatal Bereavement Scale, and the Male Introductory Information Form were completed by their husbands. The intervention group (n=38) received midwifery care based on Swanson Care Theory in addition to routine care in accordance with clinical procedures. The control group (n=38) received only routine care in accordance with the clinical procedures. For the participants in the intervention group, a practitioner's guide based on the Swanson Care Theory consisting of the stages of 'Knowing, ' 'Being together,' 'Meeting the needs,' 'Empowering' and 'Maintaining faith' was created. In this guideline, eight interviews were conducted, four face-to-face in the clinic and four by telephone after discharge. In the first interview, immediately after the woman was admitted to the clinic
  Interventions: Other: midwifery care based on swanson care theory
- Control group (No Intervention): The women and their husbands who were assigned to this group in a randomised controlled trial were interviewed after admission to the clinic and given detailed information about the study and a consent form was filled out. Women's Introductory Information Form and General Well-Being Scale Short Form, Perinatal Bereavement Scale Short Version and Male Introductory Information Form were filled out for their husbands.
  During the study period, women in this group received routine midwifery care and counselling in accordance with hospital and clinical procedures. Clinical procedures included physiological care such as bleeding control and monitoring of vital signs during termination of pregnancy. No care procedures other than physiological care were applied.
  On the thirtieth day after the woman was discharged from the clinic, the General Well-Being Scale and Perinatal Bereavement Scale were completed by telephone interview method.

INTERVENTIONS:
Other: midwifery care based on swanson care theory — All stages in the Midwifery Care and Counselling Practitioner Guide for Couples Experiencing Pregnancy Loss, which was developed by the researcher and included care, education and midwife counselling consisting of eight interviews, four of which were face-to-face and four by telephone, were applied.
  Arms: Experimental Intervention group (Group receiving midwifery care based on Swanson Care Theory)

SUMMARY:
This study was designed as a randomised controlled, 2-group, pre-test-post-test comparative, experimental study to increase the general well-being of women experiencing pregnancy loss and to decrease the level of perinatal grief.

DETAILED DESCRIPTION:
Objective: The aim of this study was to examine the effect of midwifery care and counselling based on Swanson Care Theory for couples experiencing pregnancy loss on womens perinatal grief and general well-being levels.

Method: The study had an experimental two-group pretest-posttest design. Midwifery care and counselling based on Swanson Care Theory is a grief support program consisting of eight interviews, including four face-to-face interviews after the woman's admission to the clinic and four telephone interviews until the 30th day after discharge. The study was conducted with 76 couples admitted to the obstetrics and gynecology department of a training and research hospital in Istanbul between August 2023 and May 2024 with a diagnosis of pregnancy loss. The intervention group (n=38) received midwifery care and counselling based on Swanson Care Theory in addition to routine midwifery care in accordance with clinical procedures, whereas the control group (n=38) received only routine midwifery care in accordance with clinical procedures. This study used the Women Experiencing Pregnancy Loss Introductory Information Form, Men Experiencing Pregnancy Loss Introductory Information Form, Perinatal Bereavement Scale, and General Well-Being Scale.

ELIGIBILITY:
Inclusion Criteria

* To agree to participate in the research with a partner.
* Speak and understand Turkish.
* To be 18 years of age or older.
* To be at least primary school graduate.
* Having experienced loss after spontaneous pregnancy.
* Not being diagnosed with a psychiatric illness.

Exclusion Criteria:

* Pregnancy loss due to medical termination
* Being pregnant with assisted reproductive techniques and experiencing pregnancy loss

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since pregnancy takes place in a woman's body, it was a woman-oriented study, and expectant fathers who experienced pregnancy loss were included in the supportive care for women.
Enrollment: 76 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
perinatal grief level | 30 days/1 month
  The Perinatal Grief Scale (32-item Short Version) developed by Toedter et al. consists of 32 items on a 5-point Likert scale. This scale assesses the degree of grief after perinatal loss. Each question on the scale was answered as 'Strongly agree, agree, undecided, disagree, strongly disagree. ' Active grief, hopelessness, and difficulty in coping were subscales of the scale. As the total perinatal grief score and the total score obtained from the subdimensions increased, it was determined that the grief level of the individual was higher. The total perinatal grief score obtained from the PMS was between 32-160. The Turkish validity and reliability of the scale was performed by 4 academicians in 2017 and the content validity index was found to be 0.95. In this study, the Cronbach's alpha value of the scale was 0.774.
General Well-Being Scale Short Form | 30 days later
  The short form of the General Well-being Scale was created as a result of the factor analysis studies of the shortening of the General Well-being Scale consisting of 65 items developed by Longo et al. in 2017 to determine the well-being of individuals. The General Well-Being Scale Short Form consisted of 14 items. In the five-point Likert-type scale, there are items such as Everything I do is valuable. "1" is not true at all and "5" is always true. The Turkish validity and reliability of the scale was carried out by 3 academicians in 2021, and as a result of the reliability studies, the internal consistency coefficient and construct reliability of the scale were found to be 0.84 and the two-half test correlation was 0.77. In this study, Cronbach's alpha value of the scale was 0.848.

CONTACTS AND LOCATIONS:
Overall Officials: Ayça DEMİR YILDIRIM, Phd, Study Chair — Üsküdar Üniversitesi
Locations (1):
- Üsküdar University, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
A research paper was planned to make individual participant data (IPD) available to other researchers.